CLINICAL TRIAL: NCT01094678
Title: Evaluation of the Safety and Performance of the Zilver® PTX™ Drug-Eluting Stent for Treating De Novo or Restenotic Lesions of the Above-the-knee Femoropopliteal Artery
Brief Title: Zilver® PTX™ Global Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-518; 100010 (Other: Cook)
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: Peripheral Aterial Disease (PAD); Peripheral Vascular Disease; Drug-Eluting Stent; Drug-Coated Stent; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Vascular Diseases; Cardiovascular Diseases

ARMS (1):
- Stent (Experimental)
  Interventions: Device: Zilver® PTX™ Stent

INTERVENTIONS:
Device: Zilver® PTX™ Stent — Stenting of the superfemoropopliteal artery.

SUMMARY:
The Zilver PTX Registry Study is a prospective, non-randomized, open-label, multicenter single-arm study enrolling patients in Europe, Asia, and North America with de novo or restenotic (including in-stent restenosis) lesions of the above-the-knee femoropopliteal artery (SFA). The primary endpoint of the study is event-free survival (EFS) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* stenosis of the above-the-knee femoropopliteal artery
* appropriate size and location of the lesion

Exclusion Criteria:

* pregnant or breast feeding
* failure or inability to give informed consent
* simultaneously participating in another drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2006-04; Primary Completion 2009-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Event-free Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dake, MD, Principal Investigator — Stanford University
Locations (4):
- Germany (3):
  - Heart Center Leipzig, Angiology, Leipzig
  - St. Franziskus Hospital Munster, Münster
  - Universitat Klinik Tubingen, Tübingen
- University of Roma La Sapienza, Rome, Italy

REFERENCES:
- [Derived] Dake MD, Fanelli F, Lottes AE, O'Leary EE, Reichert H, Jiang X, Fu W, Iida O, Zen K, Schermerhorn M, Zeller T, Ansel GM. Prediction Model for Freedom from TLR from a Multi-study Analysis of Long-Term Results with the Zilver PTX Drug-Eluting Peripheral Stent. Cardiovasc Intervent Radiol. 2021 Feb;44(2):196-206. doi: 10.1007/s00270-020-02648-6. Epub 2020 Oct 6. PMID 33025243
- [Derived] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Snyder SA, O'Leary EE, Tepe G, Scheinert D, Zeller T; Zilver PTX Investigators. Sustained safety and effectiveness of paclitaxel-eluting stents for femoropopliteal lesions: 2-year follow-up from the Zilver PTX randomized and single-arm clinical studies. J Am Coll Cardiol. 2013 Jun 18;61(24):2417-2427. doi: 10.1016/j.jacc.2013.03.034. Epub 2013 Apr 10. PMID 23583245
- [Derived] Zeller T, Dake MD, Tepe G, Brechtel K, Noory E, Beschorner U, Kultgen PL, Rastan A. Treatment of femoropopliteal in-stent restenosis with paclitaxel-eluting stents. JACC Cardiovasc Interv. 2013 Mar;6(3):274-81. doi: 10.1016/j.jcin.2012.12.118. PMID 23517839
- [Derived] Dake MD, Scheinert D, Tepe G, Tessarek J, Fanelli F, Bosiers M, Ruhlmann C, Kavteladze Z, Lottes AE, Ragheb AO, Zeller T; Zilver PTX Single-Arm Study Investigators. Nitinol stents with polymer-free paclitaxel coating for lesions in the superficial femoral and popliteal arteries above the knee: twelve-month safety and effectiveness results from the Zilver PTX single-arm clinical study. J Endovasc Ther. 2011 Oct;18(5):613-23. doi: 10.1583/11-3560.1. PMID 21992630